CLINICAL TRIAL: NCT04776083
Title: Role of Radiotherapy to the Primary Lesion in Metastatic Non-small Cell Lung Cancer Patients After First Line Systemic Therapy
Brief Title: Radiotherapy to the Primary in Metastatic Non-small Cell Lung Cancer Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, yostena nagy kamel mekhail, Principal Investigator, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 174 Lung Cancer
Record Dates: First submitted 2021-02-25; First posted 2021-03-01 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Non-Small Cell Carcinoma of Lung, TNM Stage 4; Radiation Therapy
Keywords: bronchogenic cancer; lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- radiotherapy arm (Experimental): after first line systemic therapy, patients will receive radiotherapy to the primary lesion, hypo-fractionated regimen 45gy will be given over 15 fractions
  Interventions: Drug: first line systemic therapy; Radiation: 3D radiotherapy or IMRT
- no intervention arm (Active Comparator): after first line systemic therapy, patients will be kept under follow up
  Interventions: Drug: first line systemic therapy

INTERVENTIONS:
Drug: first line systemic therapy — first line systemic therapy according to the genetic mutation 0f the patient
Radiation: 3D radiotherapy or IMRT — Hypo-fractionated radiotherapy to the primary lesion
  Arms: radiotherapy arm

SUMMARY:
study the effect of radiotherapy to the primary lesion after first line systemic therapy in metastatic non-small cell lung cancer patients.

DETAILED DESCRIPTION:
Metastatic non-small cell lung cancer patients after receiving their first line systemic therapy according to their genetic mutation will be randomized to follow up versus radiotherapy to the primary lesion.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed histological diagnosis of NSCLC.
2. Stage IV disease.
3. Patients with P.S ≤ 2.
4. finished at least 4 cycles of platinum-based doublet chemotherapy if patient has no diver mutation, or at least 3 months of anti-EGFR, Anti-ALK according to their driver mutation with SD, PR or CR.

Exclusion Criteria:

1. History of prior irradiation to the lung.
2. residual Malignant pleural or pericardial effusion at randomization time.
3. History of prior malignant tumor likely to interfere with the treatment protocol.
4. Severe comorbidities as measured by morbidity index.
5. Disease progression on first line systemic therapy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2020-09-25 (Actual); Primary Completion 2023-11-25 (Actual); Study Completion 2023-11-25 (Actual)

PRIMARY OUTCOMES:
progression free survival | six months
  time from randomization till disease progression
patients quality of life | six months
  using the European Organization for Research and Treatment of Cancer core quality of life questionnaire, the EORTC QLQ-C30

SECONDARY OUTCOMES:
overall survival | six months
  time from randomization till death from any cause
patients toxicity | six months
  number of participants suffer of different toxicity grades according to Common toxicity criteria of adverse events
patients pattern of failure | six months
  Number of Participants suffer of disease progression in the primary site vs other newly developed sites

CONTACTS AND LOCATIONS:
Overall Officials: Yostena Mekhail, M.Sc, Principal Investigator — Menoufia University; Eman AR Tawfeek, MD, Study Chair — Menoufia University; Enas AB Elkhouly, MD, Study Chair — Menoufia University; Reham A Abdel Aziz, MD, Study Chair — Menoufia University; Ahmed Sohaib, MD, Study Chair — Menoufia University
Locations (1):
- Medicine, Shibīn al Kawm, Menoufia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
after publishing the primary results. and if further publications will be based on these data, should add us as co investigators.
Supporting Information: Study Protocol, SAP
Time Frame: after publishing the primary results.
Access Criteria: via mail contact to the primary investigator